CLINICAL TRIAL: NCT03963349
Title: Clinical Benefit, Long Term Effectiveness, and Safety Outcome of Paroxysmal Atrial Fibrillation Ablation Using THERMOCOOL SMARTTOUCH®SF Catheters With Ablation Index
Brief Title: THERMOCOOL SMARTTOUCH®SF Catheters With Ablation Index Study
Acronym: STSF
Status: Active, not recruiting | Type: Observational
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BWI-2018-01
Record Dates: First submitted 2019-05-06; First posted 2019-05-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A single-center, real word study of consecutive subjects who undergo radiofrequency ablation for paroxysmal AF using THERMOCOOL SMARTTOUCH®SF (STSF) Catheter guiding by Ablation Index (AI). Prospectively or retrospectively record 150 eligible subjects since 1st Jan 2019 to evaluate effectiveness and safety of STSF with AI.

DETAILED DESCRIPTION:
The purpose of this study is to measure the long term effectiveness，clinical benefit, and safety outcomes of catheter ablation with STSF and AI for paroxysmal atrial fibrillation (PAF) subjects up to 12-month follow-up.

Subject:Up to 150 PAF subjects will be included in the study data, representing all consecutive subjects having catheter ablation with AI guiding STSF and for the treatment of PAF at the site.

Primary endpoint: The primary endpoint is freedom from documented atrial fibrillation (AF), atrial tachycardia (AT), or atrial flutter (AFL) (≥30 seconds) within 91-365 days post index procedure.

Secondary endpoint : Acute success at 0.5hour CPVI (i.e. entrance block achieved in all veins, verified via an isoproterenol intravenous challenge)

* Numbers of reconnected pulmonary veins (PV), with number and location of any gaps
* Procedural efficiency measures（e.g. mapping time, ablation time, total procedure time, and fluid volume delivered via catheter.
* AI values
* Inter-Tag distances
* Adverse events (Complications related to device or procedure)
* Re-hospitalization due to arrhythmia recurrence or procedure-related reasons up to 1 year Clinical Study Sites: Shanghai General Hospital Study Duration: 18-month enrollment period, with follow-up at 3, 6 and 12 months after ablation, with a blanking period defined as the period within 90 days after the ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Patient has PAF eligible for AI-guided catheter ablation with an STSF catheter per standard of care assessment
3. Able and willing to comply with all pre-, post- and follow-up testing and requirements
4. Able to sign EC-approved informed consent form

Exclusion Criteria:

1. AF is secondary to electrolyte imbalance, thyroid disease, or a reversible or non-cardiac cause
2. Patient has AF episodes lasting longer than 7 days
3. History of heart surgery, or any previous ablation for AF
4. Myocardial infarction (MI), coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI) within preceding 3 months
5. Documented left atrial thrombus on imaging
6. New York Heart Association (NYHA) class III or IV heart failure
7. Hypertrophic obstructive cardiomyopathy
8. Presence of implantable cardioverter defibrillator (ICD)
9. Contraindication to isoproterenol
10. Any other disease or malfunction that would preclude treatment with ablation in the opinion of the investigator
11. Women who are pregnant and/or breast feeding
12. Enrollment in an investigational study evaluating another device, biologic, or drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PAF population patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of freedom from documented atrial fibrillation (AF), atrial tachycardia (AT), or atrial flutter (AFL) (≥30 seconds) within 91-365 days post index procedure. | 91-365 days
  Atrial tachyarrhythmia recurrence events will be recorded and included as a study endpoint after a 90-day blanking period; recurrence during the blanking will not be considered treatment failure. In addition, re-ablation will not be recommended during the blanking period.

SECONDARY OUTCOMES:
Rate of acute success at 0.5hour CPVI | 91-365 days
  Entrance block rate achieved by all pulmonary veins after 0.5hour waiting time and isoproterenol challenge after CPVI
Numbers of reconnected pulmonary veins (PV), with number and location of any gaps | 91-365 days
  Numbers of pulmonary veins recovered after 0.5hour waiting time and isoproterenol challenge after CPVI, and the location of recovery and number are also recorded
Mapping time | 91-365 days
  Procedural efficiency measures
Contact force in grams | 91-365 days
  Ablation Index values physiological parameter of the Carto 3 which is background data generated during operation
Rate of adverse events occurred | 91-365 days
  Complications related to device or procedure
Re-hospitalization due to arrhythmia recurrence or procedure-related reasons up to 1 year | 91-365 days
  Rate of patients who are back to hospital and got hospitalized due to AF/AT/AFL recurrence or procedure-related reasons during 91 to 365 days after procedure
Ablation time | 91-365 days
  Procedural efficiency measures
Total procedure time | 91-365 days
  Procedural efficiency measures
Fluid volume delivered via catheter | 91-365 days
  Procedural efficiency measures
Ablation times in seconds | 91-365 days
  Ablation Index values physiological parameter of the Carto 3 which is background data generated during operation
Inter Tag in micrometers | 91-365 days
  Ablation Index values physiological parameter of the Carto 3 which is background data generated during operation
RF ablation and fluoroscopy times in seconds | 91-365 days
  Ablation Index values physiological parameter of the Carto 3 which is background data generated during operation

CONTACTS AND LOCATIONS:
Overall Officials: Shaowen Liu, PhD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu.